CLINICAL TRIAL: NCT01199575
Title: A Phase II Trial of Revlimid® and Rituximab, for the Treatment of Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL)
Brief Title: Phase II Trial of Revlimid® and Rituximab for Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Thomas Kipps, Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC022
Record Dates: First submitted 2010-08-31; First posted 2010-09-13 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-07

CONDITIONS: Chronic Lymphocytic Leukemia; CLL
Keywords: Chronic Lymphocytic Leukemia; CLL; Relapsed or Refractory; previously treated
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence | interventions — Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Revlimid + Rituximab (Experimental): A: Lenalidomide starting at a low dose 2.5 or 5 mg, 21 days/cycle escalated based on patient tolerability. Rituximab at 375mg/m2 administered following the first 21 days of lenalidomide monotherapy, continued weekly throughout cycle 2, and then every 4 weeks for subsequent cycles (3-7). Each patient may receive up to 7 cycles of treatment with the combination lenalidomide/rituximab if no progressive disease or significant toxicity. Patients with residual disease can elect to receive 6 additional cycles of single agent Revlimid as consolidation.
  Each patient may receive up to a maximum of 13 cycles of treatment if no progressive disease or significant toxicity.
  Interventions: Drug: Revlimid; Drug: Rituximab

INTERVENTIONS:
Drug: Revlimid
  Other Names: lenalidomide
Drug: Rituximab
  Other Names: Rituxan

SUMMARY:
The Chronic Lymphocytic Leukemia (CLL) Research Consortium (CRC) is conducting a two-arm, multi-center phase II trial of Revlimid® and rituximab for Relapsed or Refractory CLL for patients under the age of 65 and patients 65 years and older.

Lenalidomide (Revlimid) is an immunomodulatory agent with promising clinical activity in CLL and is FDA approved for treatment of relapsed multiple myeloma and 5q-myelodysplastic syndrome. Rituximab (Rituxan) is a monoclonal antibody to CD20 that is approved for the treatment of CLL.

The primary objective of this study is to determine the overall response rate of the combination of Revlimid® and rituximab in previously treated CLL patients. All patients will receive treatment with Revlimid® starting at a low dose that will be dose escalated based on individual patient tolerability. The combination of Revlimid and Rituximab will be administered for a maximum of 7 cycles. Patients with residual leukemia following seven cycles of treatment with the combination may elect to continue on protocol for an additional 6 cycles of single agent Revlimid® consolidation.

DETAILED DESCRIPTION:
The Chronic Lymphocytic Leukemia (CLL) Research Consortium (CRC) is conducting a two-arm, multicenter phase II trial of Revlimid® and rituximab for Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL) for patients under the age of 65 and patients 65 years and older.

Revlimid® (lenalidomide) a derivative of thalidomide with immune-modulating properties. Revlimid® is FDA approved for treatment of relapsed multiple myeloma and 5q- myelodysplastic syndrome. Revlimid® has promising clinical activity, in both previously treated and treatment naive CLL in early clinical trials. However, the mechanism(s) whereby Revlimid® is active in CLL is unknown. Rituximab (Rituxan®) is a monoclonal antibody that binds to CD20 expressed on normal and leukemia B cells. Rituximab is approved for the treatment of CLL.

In preclinical models of lymphoma Revlimid improved the activity of Rituximab. In clinical studies of relapsed and/or refractory CLL the combination Revlimid and Rituximab was associated with better therapeutic effects compared with what was historically observed with either agent alone.

The purpose of this study is to evaluate the safety and activity of the combination of Revlimid® and rituximab in relapsed or refractory CLL, elucidate the mechanism of action of Revlimid® in CLL, and to assess whether prognostic factors might predict those patients likely to benefit from this therapy in the future.

The primary objective of this study is to determine the overall response rate (ORR) of the combination of Revlimid® and rituximab in previously treated CLL patients for those age 65 years and above and those younger than 65.

Secondary objectives will evaluate the safety of the combination of Revlimid® and Rituximab, response duration, improvement in hematologic parameters, activity of the combination in high-risk CLL subsets, the significance of the tumor flare reaction and to compare the activity of this regimen when administered to previously treated patients to our protocol in the front line setting and to compare these outcomes for both arms of the study.

All patients will receive treatment with Revlimid® starting at a low dose that will be slowly dose escalated based on individual patient tolerability. The combination of Revlimid and Rituximab will be administered for a maximum of 7 cycles. Patients with residual leukemia following seven cycles of treatment with the combination may elect to continue on protocol for an additional 6 cycles of single agent Revlimid® consolidation.

All patients will have baseline assessment of known CLL prognostic factors through the CRC tissue core. These known prognostic features in CLL together with novel prognostic factors will be evaluated for the ability to predict response to treatment with Revlimid® and the combination of Revlimid® and Rituximab.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of chronic lymphocytic leukemia (CLL).
2. Subjects must have active disease appropriate for therapy.
3. Previous treatment for CLL
4. Understand and voluntarily sign an informed consent form.
5. Age ≥18 years at the time of signing the informed consent form.
6. Able to adhere to the study visit schedule and other protocol requirements.
7. ECOG performance status of ≤ 2 at study entry (see Appendix B).
8. Laboratory test results within these ranges: Absolute neutrophil count ≥ 1.0 x 109/L,Platelet count ≥ 50 x 109/L, Total bilirubin ≤ 1.5 mg/dL, AST (SGOT) and ALT (SGPT) ≤ 2 x ULN, Creatinine clearance estimated to be ≥ 30 ml/min
9. Disease free of prior malignancies for ≥ 2 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma in situ" of the cervix or breast.
10. Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting Revlimid® and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking Revlimid®. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. See Appendix: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods, AND also Appendix: Education and Counseling Guidance Document.

Exclusion Criteria:

1. Known Hepatitis B Ag positive, Hepatitis C positive patients.
2. Known HIV positive patients.
3. Patients with uncontrolled Autoimmune Hemolytic Anemia (AIHA) or autoimmune thrombocytopenia (ITP).
4. Inability to provide informed consent.
5. Concurrent malignancy (excluding basal and squamous cell skin cancers).
6. Active fungal, bacterial, and/or viral infection.
7. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
8. Pregnant or breast-feeding females. (Lactating females must agree not to breast feed while taking Revlimid®).
9. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
10. Use of any other experimental drug or therapy within 28 days of baseline.
11. Known hypersensitivity to thalidomide.
12. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
13. Concurrent use of other anti-cancer agents or treatments.
14. Patients with history of deep venous thrombus or pulmonary embolism. Patients who are at increased risk of thrombosis during treatment with Revlimid® including those taking concurrent erythropoietin, darbepoetin or high-dose corticosteroids are also excluded.
15. Patients with a history of embolic events (e.g. TIA) from arrhythmia or peripheral arterial disease or of recent mycocardial infarction whether or not treated with anti-platelet drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2022-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Kipps, MD, PhD, Study Director — Director of the CLL Research Consortium and University of California San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- See also: Website for the CLL Research Consortium — http://cllresearch.com/
- See also: Moore's UCSD Cancer Center — http://cancer.ucsd.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Revlimid + Rituximab: Lenalidomide starting at a low dose 2.5 or 5 mg, 21 days/cycle escalated based on patient tolerability. Rituximab at 375mg/m2 administered following the first 21 days of lenalidomide monotherapy, continued weekly throughout cycle 2, and then every 4 weeks for subsequent cycles (3-7). Each patient may receive up to 7 cycles of treatment with the combination lenalidomide/rituximab if no progressive disease or significant toxicity. Patients with residual disease can elect to receive 6 additional cycles of single agent Revlimid as consolidation.
  Each patient may receive up to a maximum of 13 cycles of treatment if no progressive disease or significant toxicity.
Period: Overall Study
Arm/Group | Revlimid + Rituximab
Started | 30
Completed | 25
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Revlimid + Rituximab
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Time Frame: nine months
Measure: Count of Participants; unit: Participants
Groups:
- Revlimid + Rituximab: A: Lenalidomide starting at a low dose 2.5 or 5 mg, 21 days/cycle escalated based on patient tolerability. Rituximab at 375mg/m2 administered following the first 21 days of lenalidomide monotherapy, continued weekly throughout cycle 2, and then every 4 weeks for subsequent cycles (3-7). Each patient may receive up to 7 cycles of treatment with the combination lenalidomide/rituximab if no progressive disease or significant toxicity. Patients with residual disease can elect to receive 6 additional cycles of single agent Revlimid as consolidation.
  Each patient may receive up to a maximum of 13 cycles of treatment if no progressive disease or significant toxicity.
  Revlimid
  Rituximab
Arm/Group | Revlimid + Rituximab
Number analyzed (Participants) | 25
Participants | 25

2. Secondary Outcome: Adverse Events to Study Treatment
Time Frame: one year
Measure: Count of Participants; unit: Participants
Arm/Group | Revlimid + Rituximab
Number analyzed (Participants) | 25
Participants | 25

3. Secondary Outcome: Progression Free Survival.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Revlimid + Rituximab
Number analyzed (Participants) | 25
Participants | 13

4. Secondary Outcome: Conversion of MRD-positive Complete Response or Partial Response (PR) to a MRD-negative Complete Response (CR) or Complete Response (CR) Respectively Following an Additional 6 Cycles of Revlimid Consolidation
Time Frame: 13 cycles
Measure: Count of Participants; unit: Participants
Arm/Group | Revlimid + Rituximab
Number analyzed (Participants) | 25
Participants | 3

5. Secondary Outcome: Overall Survival
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Revlimid + Rituximab
Number analyzed (Participants) | 25
Participants | 22

6. Secondary Outcome: Treatment Free Survival.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Revlimid + Rituximab
Number analyzed (Participants) | 25
Participants | 6

ADVERSE EVENTS:
Description: standard questionnaire, regular investigator assessment, regular laboratory testing, or other method
Arm/Group | Revlimid + Rituximab
Serious Adverse Events (participants affected / at risk) | 11/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revlimid + Rituximab (N=25)
neutropenia (Blood and lymphatic system disorders) | 7 (9)
hypophosphatemia (Blood and lymphatic system disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Bullous arthropod reaction (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revlimid + Rituximab (N=25)
abdominal distension (Gastrointestinal disorders) | 5 (6)
acid reflux (Gastrointestinal disorders) | 1 (1)
acidosis (Blood and lymphatic system disorders) | 5 (5)
acute renal failure (Renal and urinary disorders) | 1 (1)
alkaline phosphatase increase (Hepatobiliary disorders) | 7 (7)
allergic reaction (Immune system disorders) | 1 (1)
alopecia (General disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 16 (26)
anorexia (Metabolism and nutrition disorders) | 11 (14)
anxiety (Social circumstances) | 15 (29)
arthralgia (Musculoskeletal and connective tissue disorders) | 5 (8)
arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
arthritis (gout big toe) (Musculoskeletal and connective tissue disorders) | 1 (1)
atrial fibrillation (Cardiac disorders) | 2 (2)
bicarbonate decrease (Blood and lymphatic system disorders) | 1 (1)
bladder infection (Infections and infestations) | 1 (1)
bladder spasm (Renal and urinary disorders) | 1 (1)
blood biliruben increase (Blood and lymphatic system disorders) | 5 (6)
blurred vision (Eye disorders) | 1 (1)
body aches (Musculoskeletal and connective tissue disorders) | 2 (4)
bradycardia (Cardiac disorders) | 6 (8)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
bronchospasm/wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
bruising (General disorders) | 4 (5)
bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
canker sore (Skin and subcutaneous tissue disorders) | 3 (5)
chills/rigors (General disorders) | 15 (21)
cognitive disturbance (Nervous system disorders) | 1 (1)
cognitive impairment (Nervous system disorders) | 1 (1)
confusion (Nervous system disorders) | 2 (2)
conjunctivitis (Eye disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 14 (20)
cough (General disorders) | 18 (23)
cyst (Skin and subcutaneous tissue disorders) | 1 (1)
dehydration (General disorders) | 6 (7)
depression (Psychiatric disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 14 (27)
distress (Social circumstances) | 5 (5)
diverticulitis (Gastrointestinal disorders) | 1 (1)
dizziness (Nervous system disorders) | 11 (15)
dry mouth (General disorders) | 4 (4)
dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
dysesthia (Nervous system disorders) | 1 (1)
dysgeusia (Nervous system disorders) | 1 (1)
dyspepsia (Gastrointestinal disorders) | 7 (7)
dysphagia (General disorders) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
dysuria (Renal and urinary disorders) | 2 (2)
early satiety (Metabolism and nutrition disorders) | 3 (3)
ecchymosis (General disorders) | 4 (4)
edema (General disorders) | 13 (14)
edema - eyelid (General disorders) | 1 (1)
edema - facial (General disorders) | 1 (1)
elevated ALT (Hepatobiliary disorders) | 12 (15)
elevated AST (Hepatobiliary disorders) | 15 (16)
elevated creatinine (Renal and urinary disorders) | 10 (15)
elevated LDH (General disorders) | 5 (6)
elevated TSH (Endocrine disorders) | 1 (1)
epistaxis (General disorders) | 4 (4)
fatigue (General disorders) | 19 (28)
febrile illness (Infections and infestations) | 1 (1)
fever (General disorders) | 14 (18)
flatulance (Gastrointestinal disorders) | 4 (6)
fluid retention (Renal and urinary disorders) | 1 (1)
flu-like symptoms (General disorders) | 13 (19)
flushing (General disorders) | 1 (1)
fracture (Injury, poisoning and procedural complications) | 1 (1)
gait disturbance (Musculoskeletal and connective tissue disorders) | 2 (2)
gastroenteritis (Gastrointestinal disorders) | 1 (2)
general muscle weakness (Musculoskeletal and connective tissue disorders) | 12 (18)
GERD (Gastrointestinal disorders) | 1 (1)
GI Problems (Gastrointestinal disorders) | 1 (1) — Alternating constipation and diarrhea - continued through entirety of treatment.
headache (General disorders) | 8 (13)
hematoma (Blood and lymphatic system disorders) | 1 (1)
hematoma - retroperritoneal (Blood and lymphatic system disorders) | 1 (1)
hemolysis (Blood and lymphatic system disorders) | 1 (1)
hemorrhage - cut (Injury, poisoning and procedural complications) | 1 (1)
hemorrhage - oral (General disorders) | 3 (3)
hemorrhage - rectal (General disorders) | 1 (3)
high cholesterol (Blood and lymphatic system disorders) | 1 (1)
hoarseness (General disorders) | 1 (1)
hot flashes (General disorders) | 3 (6)
hydronephrosis (Renal and urinary disorders) | 1 (1)
hypercalcemia (Blood and lymphatic system disorders) | 2 (5)
hyperhidrosis (General disorders) | 14 (17)
hyperkalemia (Blood and lymphatic system disorders) | 7 (7)
hypermagnesemia (Blood and lymphatic system disorders) | 1 (1)
hypernatremia (Blood and lymphatic system disorders) | 1 (2)
hyperphosphatemia (Blood and lymphatic system disorders) | 12 (19)
hypertension (Vascular disorders) | 4 (4)
hyperuricemia (Blood and lymphatic system disorders) | 7 (15)
hypoalbuminemia (Blood and lymphatic system disorders) | 8 (9)
hypocalcemia (Blood and lymphatic system disorders) | 20 (30)
hypokalemia (Blood and lymphatic system disorders) | 3 (6)
hypomagnesemia (Blood and lymphatic system disorders) | 1 (1)
hyponatremia (Blood and lymphatic system disorders) | 15 (25)
hypophosphatemia (Blood and lymphatic system disorders) | 15 (23)
hypotension (Vascular disorders) | 8 (10)
hypothyroidism (Endocrine disorders) | 1 (2)
infusion reaction - cytokine release syndrome (Injury, poisoning and procedural complications) | 2 (2)
insomnia (General disorders) | 14 (23)
keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
keratosis - actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (2)
laryngitis (Infections and infestations) | 1 (1)
lesion (Skin and subcutaneous tissue disorders) | 5 (5)
leukopenia (Blood and lymphatic system disorders) | 1 (2)
libido decrease (General disorders) | 1 (1)
low uric acid (Blood and lymphatic system disorders) | 1 (1)
lumbar disc disease (Musculoskeletal and connective tissue disorders) | 1 (1)
memory impairment (Nervous system disorders) | 3 (3)
myalgia (Musculoskeletal and connective tissue disorders) | 14 (22)
nausea (Gastrointestinal disorders) | 16 (23)
neuropathy (Nervous system disorders) | 10 (13)
neuropathy - leg and finger spasms (Nervous system disorders) | 1 (1)
neutropenia (Blood and lymphatic system disorders) | 22 (42)
night sweats (General disorders) | 14 (20)
osteopenia (Musculoskeletal and connective tissue disorders) | 2 (2)
pain - abdominal (General disorders) | 10 (14)
pain - abdominal/stomach - cramps (Musculoskeletal and connective tissue disorders) | 1 (3)
pain - back (General disorders) | 11 (18)
pain - chest (General disorders) | 4 (5)
pain - chest - non-cardiac (General disorders) | 1 (1)
pain - ear (General disorders) | 2 (2)
pain - extremity (General disorders) | 14 (19)
pain - eye (General disorders) | 1 (1)
pain - facial (General disorders) | 1 (2)
pain - hip (General disorders) | 4 (6)
pain - knee (General disorders) | 1 (1)
pain - lymph node (General disorders) | 3 (3)
pain - neck (General disorders) | 2 (3)
pain - pharyngolaryngeal (General disorders) | 12 (14)
pain - rectal (General disorders) | 1 (1)
pain - ribs (General disorders) | 1 (2)
pain - right disessciata (General disorders) | 1 (1)
pain - right side (General disorders) | 1 (1)
pain - skin (Nervous system disorders) | 1 (1)
pain - stomach (General disorders) | 9 (12)
pain - tumor (General disorders) | 12 (16)
palmar-plantar erythrodysesthia (Injury, poisoning and procedural complications) | 1 (1) — Treatment reaction
palpitations (Cardiac disorders) | 2 (2)
prostatitis (Reproductive system and breast disorders) | 2 (2)
proteinuria (Renal and urinary disorders) | 1 (1)
pruritis (Skin and subcutaneous tissue disorders) | 10 (16)
psychosis (Psychiatric disorders) | 1 (1)
purpura (Vascular disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 15 (24)
restless leg syndrome (General disorders) | 1 (1)
retinal detachment (Eye disorders) | 1 (1)
rhinitis (General disorders) | 2 (2)
rhinitis - allergic rhinitis (Immune system disorders) | 11 (16)
right eye floater (Eye disorders) | 1 (1)
sciatica (Nervous system disorders) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
sinus arrhythmia (Cardiac disorders) | 1 (1)
sinusitis (Infections and infestations) | 5 (8)
skin and subcutaneous tissue disorder (Skin and subcutaneous tissue disorders) | 1 (1)
skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 5 (5)
skin infection (Skin and subcutaneous tissue disorders) | 2 (2)
skin infection - cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
skin ulceration (Skin and subcutaneous tissue disorders) | 3 (4)
skin ulceration - blister on roof of mouth (Skin and subcutaneous tissue disorders) | 1 (1)
skin ulceration - finger (Skin and subcutaneous tissue disorders) | 1 (1)
small intestine infection (Gastrointestinal disorders) | 1 (1)
superficial phlebitis (Vascular disorders) | 1 (1)
swelling - tongue (General disorders) | 1 (1)
syncope (General disorders) | 2 (2)
tachycardia (Cardiac disorders) | 3 (3)
taste alteration (Nervous system disorders) | 1 (1)
tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2)
thrombocytopenia (Blood and lymphatic system disorders) | 20 (28)
thrombophlebitis (Vascular disorders) | 1 (1)
thrombophlebitis - superficial (Vascular disorders) | 4 (7)
tinnitus (Ear and labyrinth disorders) | 1 (1)
tremors (Nervous system disorders) | 3 (3)
tumor flare reaction (Injury, poisoning and procedural complications) | 3 (5) — Treatment reaction
ulcer - mouth (Skin and subcutaneous tissue disorders) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 13 (16)
urinary frequency (Renal and urinary disorders) | 10 (12)
urinary retention (Renal and urinary disorders) | 2 (2)
urinary tract infection (Renal and urinary disorders) | 2 (2)
urine discoloration (Renal and urinary disorders) | 2 (2)
urine odor (Renal and urinary disorders) | 1 (1)
urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
vaginal odor (Reproductive system and breast disorders) | 1 (1)
ventricular arrhythmia (Cardiac disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 8 (9)
watering eyes (Eye disorders) | 1 (1)
weight gain (Metabolism and nutrition disorders) | 1 (1)
weight loss (Metabolism and nutrition disorders) | 15 (18)
yeast (vaginal) infection (Reproductive system and breast disorders) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes